CLINICAL TRIAL: NCT00202280
Title: VIP (Vitamins In Psychosis) Study. A Randomized Double Blind Placebo Controlled Trial of the Effects of Vitamin B12, B6 and Folic Acid Augmentation on Cognition and Symptoms in Early Psychosis.
Brief Title: Efficacy of Treating First Episode Psychosis With Folic Acid,B12 and B6 in Addition to Antipsychotic Medication
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Melbourne Health (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPREC 26/2004; 03T-472 (Other Grant/Funding Number: Stanley Medical Research Institute)
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: First Episode Psychosis
MeSH Terms: interventions — Folic Acid; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo pill (Placebo Comparator): Placebo pill daily for 3 months
  Interventions: Drug: Folic Acid 5mg, Vitamin B12 0.4mg and B6 50mg
- 5mg folic acid, 0.4mg B12, 50mg B6 (Experimental): 5mg folic acid, 0.4mg B12, 50mg B6 in one pill, daily for 3 months
  Interventions: Drug: Folic Acid 5mg, Vitamin B12 0.4mg and B6 50mg

INTERVENTIONS:
Drug: Folic Acid 5mg, Vitamin B12 0.4mg and B6 50mg

SUMMARY:
The purpose of this study is to determine whether Vitamin B12,B6 and Folic Acid are effective with antipsychotic medication in the treatment of First Episode Psychosis.The B-complex Vitamins' homocysteine lowering properties may have an effect on cognition and symptoms. We are examining changes in symptoms and cognition over a 3 month period.

DETAILED DESCRIPTION:
The core rationale of this study will be to prospectively investigate whether Vitamin B12, B6 and Folic Acid and the associated lowering of homocysteine levels will improve and /or protect cognitive functioning in a cohort of 120 first episode psychosis patients.

This is a randomized, double blind placebo controlled add on standard therapy trial with vitamin B12, B6 and folic acid, in young patients between 15-25 presenting to ORYGEN Youth Health with a first psychotic episode . Vitamins (B12 , B6 and Folate) will be compared with placebo added to standard treatment for a period of 12 weeks in a double blind fashion. Primary outcome measures will be psychopathology and cognition (CogState and MATRICS). Secondary outcome measures will be tolerability and safety measures (drop-out rates, general side effect scale (UKU).

Patients who give informed consent will be randomised to receive treatment with vitamin (5 mg folic acid, 0.4 mg B12, and 50 mg B6) daily or placebo for 12 weeks.

Patients will be randomised by a dynamic randomisation method called minimization which allocates patients to treatment group by checking the allocation of similar patients already randomised, and allocating the next treatment group "live" to best balance the treatment groups across all stratification variables. The minimization will be carried out by the NHMRC clinical trials centre in Sydney , and the patient will be randomized to either placebo or vitamin. Each patient will collect their tablets from the clinical trials pharmacy. The Clinical Trials Pharmacy will dispense either vitamin or placebo. All study personnel and participants will be blinded to treatment assignment for the duration of the study. To enhance the quality of measurement (and increase the power of the study by avoiding dilution of effect) adherence to medication will be measured electronically with electronic pill caps (Medication Event Monitoring System VI, ARRDEX Ltd). This will allow us to assess actual pharmacological exposure in an objective manner.

ELIGIBILITY:
Inclusion Criteria:

* Male and females
* Between 15 and 25 years of age
* First Episode Psychosis
* 3 months of treatment
* Attending ORYGEN Youth Health, a geographical based catchment area service for young people aged between 15 and 25

Exclusion Criteria:

* Untreated B12 deficiency or untreated pernicious anaemia
* Patients on multi-vitamins, single B6, or folic acid, unless willing to discontinue and take study supplement
* Chronic haemolytic states such as thalassaemia major or sickle-cell anaemia
* Hypersensitivity to folic acid
* Organic disorders presenting with a psychotic syndrome (e.g. brain tumour, temporal lobe epilepsy, HIV encephalopathy)
* Mental retardation (unable and/or unlikely to give appropriate information of symptomatology or side-effects (IQ approximately lower than 70)
* History of clinically significant physical illness (e.g. terminal cancer, renal dialysis)
* History of brain surgery
* History of brain infarction
* Pregnant or lactating women, or women of childbearing potential not using an acceptable method of contraception

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2004-09; Primary Completion 2006-09 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Cognition (MATRICS and COGSTATE)at 3 months
Symptomatology at 3 months

SECONDARY OUTCOMES:
Safety at 3 months
Tolerability at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Colin P O'Donnell, MB,MRCPsych, Principal Investigator — ORYGEN Research Centre , ORYGEN Youth Health,Department of Psychiatry, University of Melbourne; Prof Patrick D McGorry, PhD FRANZP, Study Director — ORYGEN Research Centre , ORYGEN Youth Health,Department of Psychiatry, University of Melbourne
Locations (1):
- ORYGEN Youth Health, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Allott K, McGorry PD, Yuen HP, Firth J, Proffitt TM, Berger G, Maruff P, O'Regan MK, Papas A, Stephens TCB, O'Donnell CP. The Vitamins in Psychosis Study: A Randomized, Double-Blind, Placebo-Controlled Trial of the Effects of Vitamins B12, B6, and Folic Acid on Symptoms and Neurocognition in First-Episode Psychosis. Biol Psychiatry. 2019 Jul 1;86(1):35-44. doi: 10.1016/j.biopsych.2018.12.018. Epub 2019 Jan 9. PMID 30771856